CLINICAL TRIAL: NCT03761628
Title: An Open-label Study to Evaluate Clinical Performance of Gedea Pessary in Adult Women With Vulvovaginal Candidiasis
Brief Title: Clinical Performance of a Vaginal Pessary (pHyph) in Vulvovaginal Candidiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gedea Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QRS-CL1-003
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Vulvovaginal Candidiasis
Keywords: Vaginal Yeast Infection; Candidiasis, vulvovaginal; Genital diseases, female; Vaginitis; Vulvovaginitis; Vaginal diseases
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Genital Diseases, Female; Vaginitis; Vulvovaginitis; Vaginal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pHyph, Gedea Pessary (Experimental): Clinical performance, tolerability, safety and user experience of Gedea Pessary, a slow-release vaginal tablet for the treatment of VVC.
  Interventions: Device: pHyph generation I

INTERVENTIONS:
Device: pHyph generation I — A vaginal tablet for the treatment of VVC to be administered every 48 hours
  Other Names: Gedea pessary

SUMMARY:
This is an open-label, single-armed, multi-center study to evaluate clinical performance, tolerability, and safety of Gedea Pessary in 24 adult women with vulvovaginal candidias (VVC). On Day 0, patients will have gynecological examination, vaginal samples taken, and will receive the investigational product to be self-administered. Patients will be examined after 7 days with respect to VVC signs and symptoms and if not cured, will receive prolonged treatment for one additional week. Patients will be followed-up by telephone up to 29 days after last treatment. Vaginal samples will be used for confirming diagnosis and microbiome analyzes. Patient questionnaires will be used for assessing VVC symptoms, usability, and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Adult, post-menarchal, pre-menopausal women aged 18 years or older
* Diagnosis of VVC, defined as having a white or creamy vaginal discharge plus the following findings:

  1. At least 2 of the following signs and symptoms of VVC that are characterized as at least moderate: itching, burning, irritation, edema, redness, or excoriation.
  2. Potassium hydroxide (KOH) or saline preparation from the inflamed vaginal mucosa or secretions revealing yeast forms (hyphae or pseudohyphae) or budding yeasts.
* Having decisional capacity and providing written informed consent
* Negative urine pregnancy test at screening
* Refrain from using any intravaginal products (i.e., contraceptive creams, gels, foams, sponges, lubricants, or tampons, etc.) during the study period
* Refrain from sexual intercourse or use a condom until Day 7
* Signed informed consent and willing and able to comply with all study requirements

Exclusion Criteria:

* Patients with known or apparent signs of other infectious causes of VVC (BV, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, Herpes simplex, or human papillomavirus) at screening
* Patients who are pregnant or breastfeeding
* Patients who were treated for VVC within the past 14 days
* Patients who are currently receiving antifungal therapy unrelated to VVC or has taken antifungal therapy within the past 14 days
* Patients who have used pH-modifying vaginal products within the last 14 days
* Patients who have received an investigational drug in a clinical investigation within 30 days prior to screening
* Known/previous allergy or hypersensitivity to any product constituent or fluconazole
* Any medical condition that in the Investigator's judgments would make the patient unsuitable for inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Cardell, MD, PhD, Principal Investigator — Kvinnokliniken, Region Skåne
Locations (2):
- Sweden (2):
  - Hoftekliniken, Helsingborg
  - Annerokliniken, Hofterup

REFERENCES:
- See also: Sponsor webpage — http://gedeabiotech.com

RESULTS

PARTICIPANT FLOW:
Groups:
- pHyph, Gedea Pessary: Clinical performance, tolerability, safety and user experience of Gedea Pessary, a slow-release vaginal tablet for the treatment of VVC.
  pHyph, Gedea pessary: pHyph is a vaginal tablet for the treatment of VVC
Period: Overall Study
Arm/Group | pHyph, Gedea Pessary
Started | 23 (Received study treatment)
Completed | 17
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: A total of 24 participants were enrolled, whereof 23 participants received study treatment.
Groups:
- pHyph, Gedea Pessary: Clinical performance, tolerability, safety and user experience of Gedea Pessary, a slow-release vaginal tablet for the treatment of vulvovaginal candidiasis (VVC).
  pHyph, Gedea pessary: pHyph is a vaginal tablet for the treatment of VVC
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 23
Experience of any vaginal candida infection during the last 12 months [Count of Participants; unit: Participants]
  Yes | 22
  No | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate
Description: Clinical cure was defined as the absence of signs and symptoms of vulvovaginal candidiasis (VVC) in terms of having a composite vulvovaginal signs-and-symptoms (CVVS) score equal to or below 3.
  * Each of the following 6 vulvovaginal signs and symptoms were individually scored using the scoring scale below and then added together to determine the CVVS score.
    * Vulvovaginal signs: erythema, edema, or excoriation
    * Vulvovaginal symptoms: itching, burning, or irritation
  * Scoring Scale: each score should be objectively defined. 0 = none (absent)
    1. = mild (slight)
    2. = moderate (definitely present)
    3. = severe (marked, intense)
Time Frame: Day 7
Population: The Full analysis set population contained 23 patients. One patient was not included in this analysis due to missing clinical cure data (CVVS score).
Measure: Count of Participants; unit: Participants
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 22
Participants | 9
Statistical Analysis 1: Comparison: pHyph, Gedea Pessary; It was assumed that the true cure rate was equal to 70%, therefore 22 patients were needed to obtain 90% chance (90% power) to show that the one-sided 95% CI for the observed cure rate was above 40%. Hypotheses for the primary clinical performance endpoint: * Null hypothesis: Clinical cure rate is less than or equal to 40%. * Alternative hypothesis (one-sided): Clinical cure rate is above 40%; Test type: Other — The clinical performance endpoint - Clinical cure rate on Day 7 - was calculated and presented together with a one-sided 95% CI based on the exact binomial distribution (Clopper-Pearson); Clinical cure rate = 40.9, 95% CI 1-sided [lower limit 23.3]

2. Secondary Outcome: Proportion of Patients Having a Reduction in CVVS Score
Description: Defined as the absence of signs and symptoms of vulvovaginal candidiasis (VVC) in terms of having a composite vulvovaginal signs-and-symptoms (CVVS) score equal to or below 3.
  - Each of the following 6 vulvovaginal signs and symptoms were individually scored using the scoring scale below and then added together to determine the CVVS score.
  * Vulvovaginal signs: erythema, edema, or excoriation
  * Vulvovaginal symptoms: itching, burning, or irritation -Scoring Scale: each score should be objectively defined: 0 = none (absent)
    1. = mild (slight)
    2. = moderate (definitely present)
    3. = severe (marked, intense)
Time Frame: Day 7 compared to Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 22
Participants | 16
Statistical Analysis 1: Comparison: pHyph, Gedea Pessary; Test type: Other — Results are based on the exact binomial distribution (Clopper-Pearson); Proportion with reduction = 72.7, 95% CI 2-sided [49.8 to 89.3]

3. Secondary Outcome: Usability, Measured by Patient Questionnaire
Description: General assessment of the treatment on a integer scale that ranges from 1 to 10. The lower end of the scale is indicated with the term "Not satisfied" and the higher end with the term "Very satisfied".
  Question asked: How do you generally regard the treatment?
Time Frame: Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Integer scale (1-10)
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 22
Integer scale (1-10) | 6.4 (2.2)

4. Secondary Outcome: Proportion of Patients Having a Recurrence
Description: Proportion of patients answering [Yes] to the question "Have the symptoms recurred?"
Time Frame: Up to day 35
Population: The Full analysis set population contained 23 patients.The sub-set of the Full analysis set including patients not receiving prolonged treatment contained 9 patients. Of these, 8 patients were included in this analysis of recurrence at Day 14 and 6 patients were included in the analysis of recurrence at Day 35.
Measure: Count of Participants; unit: Participants
Arm/Group | pHyph, Gedea Pessary
Number analyzed (Participants) | 8
Participants
  Day 14 | 1
  Day 35: number analyzed (Participants) | 6
  Day 35 | 0
Statistical Analysis 1: Comparison: pHyph, Gedea Pessary; Test type: Other — Results are based on the exact binomial distribution (Clopper-Pearson); Recurrence rate Day 14 = 12.5, 95% CI 2-sided [0.3 to 52.7]
Statistical Analysis 2: Comparison: pHyph, Gedea Pessary; Test type: Other — Results are based on the exact binomial distribution (Clopper-Pearson); Recurrence rate Day 35 = 0, 95% CI 2-sided [0 to 45.9]

ADVERSE EVENTS:
Time Frame: Up to day 42
Arm/Group | pHyph, Gedea Pessary
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 12/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | pHyph, Gedea Pessary (N=23)
Headache (Nervous system disorders) | 5 (6)
Dysmenorrhoea (Reproductive system and breast disorders) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03761628/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT03761628/SAP_001.pdf